CLINICAL TRIAL: NCT07296055
Title: Evaluating the Utility of Endobronchial Valves in the Management of Tubercular and NTM (Non Tubercolar Micobacteriosis) Pulmonary Cavities
Brief Title: Endobronchial Valve in Tubercular and NTM Pulmonary Cavities.
Acronym: TBET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26268_spe; 25-01-050896 (Other: Ministry of Health)
Record Dates: First submitted 2025-12-03; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Multidrug Resistance Tubercolosis; Non Tubercolar Micobacteriosis
Keywords: Endobronchial valves; Non Tubercolar Micobacteriosis; Multidrug Resistance Tubercolosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Zephyr ® (Experimental): Patients will be randomized in the two arms. All patients will continue antibiotic therapy as per clinical practice. Within 30 days the patients allocated to the experimental arm will be contacted to schedule bronchoscopy for valve placement. The treatment will be performed on a day hospital basis, patients will undergo Chest X-rays before discharge in order to confirm correct valve placement. After 9 month the experimental arm will undergone a procedure in order to remove valves.
  Interventions: Device: Endobronchial valves
- Control (No Intervention): Patients randomized in control arm will continue antibiotic therapy as per clinical practice.

INTERVENTIONS:
Device: Endobronchial valves — Patients shall undergo a bronchoscopy in sedation using midazolam and/or fentanyl or general anaesthesia with propofol in some cases. For MDR - TB patients the procedure will be done in an isolation room with negative pressure. Rigid bronchoscopy, facial or laryngeal mask airway shall be employed to introduce the fiberoptic bronchoscope, an instrument equipped with an operating channel of variable diameter between 2.8 and 3.2 mm that allows insertion of the valve.
  The Zephyr ® EBV is a self-expandable system which is actuated to contact with the bronchial wall, facilitating adhesion to the bronchial wall and moulding in conformity with the bronchial anatomy. Being one-way valves, that prevent the ingress of the air to the segment or lobe under consideration, while allowing, egress of the same during exhalation.
  Other Names: no interventions
  Arms: Zephyr ®

SUMMARY:
Tuberculosis (TB) is a complex disease in which the lungs are the primary site of infection. Infection is acquired through inhalation of droplet nuclei laden with Mycobacterium bacilli (M. tuberculosis) that settle in the alveoli as the primary focus. TB is characterized by a gradual expansion of infection and cavitation that causes progressive tissue destruction. Furthermore, the increase in drug-resistant forms of TB, including multidrug resistance (MDR) and pre-extensively drug-resistant TB (XDR), is becoming increasingly concerning. Treatment of pharmacosensitive diseases involves a duration of no less than 6 months, while that of MDR-TB and XDR-TB are even longer; generally well above 24 months. Nontuberculous mycobacteria (NTMs), or atypical mycobacteria, are organisms that cause various diseases such as skin and soft tissue infections, lymphadenitis, lung infections, disseminated infections, and a wide range of more rarely encountered infections that do not differ from tuberculosis in anatomy and radiologically even though they usually do not develop the primary complex. Given that the treatment success rate is unsatisfactory, there is an urgent need for new drugs and additional interventions to improve outcomes, both in patients with MDR/XDR-TB and in patients with difficult-to-treat NTM.

One-way endobronchial valves (EBVs) have been used as an effective lung volume reduction strategy in emphysema without significant adverse events. The mechanism consists in inducing atelectasis, that is, creating a poorly ventilated environment with reduced oxygen tension. This reduced oxygen tension is unfavorable for the survival and proliferation of mycobacteria. Therefore, using these devices to treat cavities caused by multidrug-resistant mycobacteria or in patients not eligible for surgical therapy should reduce or completely heal the cavity, creating an inhospitable environment for the bacteria, slowing or eliminating their growth.

Condition/disease: Pulmonary MDR/XDR-TB or NTM (difficult to treat or resistant to treatment) Number of patients to be enrolled: 30 It is a single-center, randomized, controlled, open-label, two-arm study.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years AND
2. Patient with cavities deemed unsuitable for surgery (when an extensive pulmonary parenchymal damage due to TB, is present, making patients inappropriate for open thoracic surgery) AND
3. To have signed the informed consent

   AND one of the following conditions:
4. Pulmonary MDR/XDR -TB or NTM (difficult to treat or resistant to treatment) confirmed by smear samples and antibiogram or with persistence of positivity for Mycobacterium of the smear after standard pharmacotherapy and severe destruction of the lungs with 1 or more persistent cavities.
5. Pulmonary TB or NTM with cavities and associated systemic diseases such as pancreatic diabetes, stomach and duodenum ulcer, liver and kidney diseases, HIV or another such disease that compromises pharmacological treatment.
6. Recurrent haemoptysis attributable to TB or NTM

Exclusion Criteria:

1. Contraindication to performance of bronchoscopy
2. Severe cardiac comorbidities
3. Severe psychiatric disorders
4. Functional or anatomical pneumonectomy
5. Asthma
6. Pregnancy
7. Patients for whom bronchoscopic procedures are contraindicated
8. Patients with known allergies to Nitinol (nickel-titanium) or its constituent metals (nickel or titanium)
9. Patients with known allergies to silicone
10. Patients who have not quit smoking
11. Patients with large bullae encompassing greater than 30% of either lung
12. Patients with active pulmonary infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2028-05-12 (Estimated); Study Completion 2028-12-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with cavities reduction equal or above 50% in the two arms | At 9 months after the randomization
  Percentage of patients with cavity dimension, at 9 months of treatment, < or = to 50% of cavity dimension at baseline. The results will be expressed in mm, through the maximum axial diameter. Higher percentage in the experimetal arm Zephyr suggests the efficacy of the treatment.
Percentage of patients with sputum smear negative for microbiological agents in the two arms at 9 months of treatment | 9 months after the randomization
  The sputum smear for microbiological agents will be collected on a slide and then observed through optical microscopy. The results will be expressed in dichotomous scale. Higher percentage of negative results in the experimental arm Zephyr suggests the efficacy of the treatment.

SECONDARY OUTCOMES:
Median of cavity dimension differences at each timepoints in comparison with baseline in both arms. | At 3 months and 9 months after the randomization
  The difference of cavity assial diameter, expressed in mm, between each timepoints and baseline. Differences will be expressed in median and in interquartile range in each arm.
Percentage of patients with sputum smear negative for microbiological agents in the two arms, at each timepoints | At 1, 3, 9 months after randomization and at 12, 14 months at the follow up
  The sputum smear for microbiological agents will be collected on a slide and then observed through optical microscopy. The results will be expressed in semiquantitative scale. Higher percentage of negative results in the experimental arm Zephyr suggests the efficacy of the treatment.
Percentage of culture negative for microbiological agents at each timepoint among the two arms. | At 1, 3, 9 months after the randomization and 12, 14 months at the follow up
  At each timepoints sputum will be collected and cultered. The culture will be observed through optical microscopy for 8 weeks. If after 8 weeks no microbacterial growth will be observed, the negativity will be diagnosed for that sample. The results wil be expressed in CFU.
Percentage of patients with early (within 48 hours) and late complications in the experimental arm Zephyr. | At T0 (intervention)+48 hours, 3 and 9 months after intervention.
  In the experimental arm Zephyr the complications that arise within 48 hours are defined early, events after 48 hours, will be defined late complications. The severity of the complication will be assessed by CTCAE v4.0.
Percentage of patients who have undergone valve reposition in experimental arm Zephyr. | At 3 months after the intervention.
  At 3 months after intervention, the correct valve position will be confirmed through CT scan. The results will be expressed as the proportion between patients that undergone for the valve reposition and total patients evaluated at 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Careggi, Florence, FI, Italy

IPD SHARING:
Plan to Share IPD: No